CLINICAL TRIAL: NCT05107362
Title: Clinical Performance of the Checkable Medical At-Home Strep A Test
Status: Completed | Type: Observational
Sponsor: Checkable Medical Inc (Industry)
Collaborators: Curebase Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CM-003
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-03

CONDITIONS: Streptococcus Pyogenes Infection; Pharyngitis; Respiratory Tract Infections
Keywords: In vitro diagnostic
MeSH Terms: conditions — Streptococcal Infections; Pharyngitis; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Symptomatic Adult and Pediatric Subjects: Untrained lay user to collect throat swab specimen and perform investigational test.
  Interventions: Diagnostic Test: untrained lay user performs investigational diagnostic test

INTERVENTIONS:
Diagnostic Test: untrained lay user performs investigational diagnostic test — Untrained lay users (parents/guardians of pediatric subjects or friends/family members of adult subjects) collect throat swab specimens and perform the investigational diagnostic test.

SUMMARY:
The Checkable Medical At-Home Strep A Test is a rapid chromatographic immunoassay for the qualitative detection of Group A Strep (GAS) antigens from throat swabs. The purpose of the study is to evaluate the clinical performance of the investigational device (i.e., sensitivity, specificity, NPV and PPV) when used by untrained lay persons to detect the presence of Group A Streptococcal antigens in throat swab specimens from individuals five years of age and older with signs and symptoms of pharyngitis, such as fever and sore throat.

DETAILED DESCRIPTION:
The study is a prospective, consecutive, non-interventional multicenter study to evaluate the clinical performance of the Checkable Medical At-Home Strep A Test when the test is performed by non-trained adult lay users.

1. Patients or parents/legal guardians of patients presenting with signs and symptoms of pharyngeal GAS infections will be recruited at primary care or urgent care clinics.
2. Informed consent will be obtained from adult subjects and from the parents/guardians of pediatric subjects. Pediatric subjects 7 years of age or greater will be asked for their assent.
3. The lay user will be provided with a Checkable Medical At-Home Strep A Test kit. The user and patient will be provided with a quiet, private space where the user can collect the throat swab specimen and perform the investigational test.
4. Once the lay user has collected the swab sample for the Checkable Medical At-Home Strep A Test and performed the test, she/he will document the test result. The Checkable Medical At-Home Strep A Test result is not to be shared with members of the site team who are providing healthcare to the subject.
5. When all sample collection, testing and interpretation activities related to the investigational test are completed, a healthcare provider at the study site will collect two additional swab samples. One of these samples will be sent to a central lab where it will be cultured for GAS. An additional sample will be tested using the organization's standard of care (SOC) rapid Strep A test.
6. Subjects will be diagnosed and treated in accordance with routine SOC which may include an FDA-cleared rapid GAS test. The Checkable Medical At-Home Strep A Test will not be used to diagnose or treat study subjects.
7. This study will take place in at least six sites in at least three different regions of the United States.
8. The results from the Checkable Medical At-Home Strep A Test will be used to compare with the diagnostic truth obtained through culture to compute diagnostic accuracy parameters including sensitivity, NPV, specificity and PPV.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects seeking medical care for two or more of the following signs/symptoms of pharyngeal streptococcal infections:

   * pharyngeal pain [with or without swallowing],
   * tonsillar swelling with exudates,
   * pharyngeal erythema,
   * tender cervical lymphadenopathy,
   * fever.
2. Subjects who have not received antibiotic treatment within the past 14 days.
3. Subjects (or their parents/guardians) provide written informed consent/assent to participate in the study

Exclusion Criteria:

1. Lay users who are accompanying patients are unwilling/unable to collect throat swab sample from a child or adult.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 610 to 1,220 male and female subjects in the US, with approximately 183 subjects being strep positive, are expected to participate in the study. At least half of the subjects will be between 5 and 17 years of age and the remaining subjects will be adults 18 years of age and older.
Sampling Method: Non-Probability Sample
Enrollment: 1347 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Clinical Sensitivity and Clinical Specificity | 1 day
  Sensitivity is the proportion of subjects with a positive bacterial culture that are also positive in the investigational Strep A test (+).
  Specificity is the proportion of subjects with a negative bacterial culture that are also negative in the investigational Strep A test (-).

SECONDARY OUTCOMES:
Negative Predictive Value | 1 day
  Negative Predictive Value (NPV) is the proportion of subjects with negative investigational Strep A test results who also have negative cultures (diagnostic truth); calculated as 100 x d/(c+d).

CONTACTS AND LOCATIONS:
Overall Officials: Marla McIntyre, Study Director — Checkable Medical
Locations (22):
- United States (22):
  - Robertson Pediatrics, Beverly Hills, California
  - Angel Kids Pediatrics, Jacksonville, Florida
  - L&A Morales Health Care, Miami, Florida
  - Elite Clinical Trials, Blackfoot, Idaho
  - Waggoner Pediatrics, Clive, Iowa
  - WellNow Urgent Care and Research, Kalamazoo, Michigan
  - Axis Clinicals, Dilworth, Minnesota
  - Infinitive Bio Research, Edison, New Jersey
  - Twelve Corners Pediatrics, Rochester, New York
  - AFC Urgent Care, The Bronx, New York
  - Plains Clinical Research, Fargo, North Dakota
  - Trinity Health, Minot, North Dakota
  - WellNow Urgent Care and Research, Lorain, Ohio
  - WellNow Urgent Care and Research, Milford, Ohio
  - WellNow Urgent Care and Research, Troy, Ohio
  - AFC Urgent Care, Easley, South Carolina
  - Tribe Clinical Research, Greenville, South Carolina
  - MDFirst, Lancaster, South Carolina
  - Pediatric Associates, Houston, Texas
  - Santa Clara Family Clinic, Houston, Texas
  - Pediatric Center, Richmond, Texas
  - North Houston Internal Medicine and Pediatric Clinic, Tomball, Texas

IPD SHARING:
Plan to Share IPD: No